CLINICAL TRIAL: NCT00074438
Title: Randomized, Multifactorial, Double-blind, Parallel-group, Dose-ranging Study of the Efficacy and Safety of Rituximab (MabThera®/Rituxan®) in Combination With Methotrexate in Patients With Active Rheumatoid Arthritis
Brief Title: Study to Assess the Efficacy and Safety of Rituximab in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA17043/U2644g; WA17043
Record Dates: First submitted 2003-12-12; First posted 2003-12-15 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rituxan; RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Rituximab; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (9):
- 1 (Experimental)
  Interventions: Drug: methotrexate; Drug: rituximab
- 2 (Experimental)
  Interventions: Drug: methotrexate; Drug: rituximab; Drug: corticosteroids
- 3 (Experimental)
  Interventions: Drug: methotrexate; Drug: rituximab; Drug: corticosteroids
- 4 (Experimental)
  Interventions: Drug: methotrexate; Drug: rituximab
- 5 (Experimental)
  Interventions: Drug: methotrexate; Drug: rituximab; Drug: corticosteroids
- 6 (Experimental)
  Interventions: Drug: methotrexate; Drug: rituximab; Drug: corticosteroids
- 7 (Placebo Comparator)
  Interventions: Drug: methotrexate; Drug: placebo
- 8 (Placebo Comparator)
  Interventions: Drug: methotrexate; Drug: corticosteroids; Drug: placebo
- 9 (Placebo Comparator)
  Interventions: Drug: methotrexate; Drug: corticosteroids; Drug: placebo

INTERVENTIONS:
Drug: methotrexate — Oral or parenteral repeating dose
Drug: rituximab — Intravenous repeating dose
  Arms: 1; 2; 3; 4; 5; 6
Drug: corticosteroids — Intravenous repeating dose
  Arms: 2; 3; 5; 6; 8; 9
Drug: placebo — Intravenous repeating dose
  Arms: 7; 8; 9

SUMMARY:
This study will assess the efficacy and safety of different treatment regimens of rituximab (MabThera®/Rituxan®), corticosteroids, and placebo, combined with methotrexate (MTX), in patients with active rheumatoid arthritis (RA).

ELIGIBILITY:
Eligibility criteria include, but are not limited to the following:

* Are between the ages of 18 and 80 years.
* Have been diagnosed with rheumatoid arthritis for at least 6 months.
* Have failed treatment (lack of efficacy) with at least 1 but no more than 5 disease-modifying anti-rheumatic drugs or biologics (other than methotrexate).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2003-06; Primary Completion 2004-09 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with an ACR20 response | 24 weeks

SECONDARY OUTCOMES:
Proportion of patients with ACR(50,70) responses | 24 weeks
Proportion of patients with an ACR20 response in the medium- and high-dose corticosteroid groups | 24 weeks

REFERENCES:
- [Derived] Keystone E, Fleischmann R, Emery P, Furst DE, van Vollenhoven R, Bathon J, Dougados M, Baldassare A, Ferraccioli G, Chubick A, Udell J, Cravets MW, Agarwal S, Cooper S, Magrini F. Safety and efficacy of additional courses of rituximab in patients with active rheumatoid arthritis: an open-label extension analysis. Arthritis Rheum. 2007 Dec;56(12):3896-908. doi: 10.1002/art.23059. PMID 18050221